CLINICAL TRIAL: NCT02481063
Title: Differences in Muscle (Vastus Laterals and Gastrocnemius Medialis) and Tendon Adaptation (Patellar and Achilles) in Lower Extremity After 3 Running Days With a Group Trained by Eccentric Overload, Measured by Ultrasound and Thermography
Brief Title: Adaptation in Lower Extremity After 3 Running Days, With a Group Trained by Eccentric Overload
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Collaborators: University of Jaén (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: TF_US20015
Record Dates: First submitted 2015-05-27; First posted 2015-06-25 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-06

CONDITIONS: Sports Injuries
Keywords: Eccentric; Running; Muscle; Tendon; Ultrasound; Thermography
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eccentric (Active Comparator): 6 Weeks Training with eccentric Overload (Squat with Yoyo Technology) 3 Consecutive Days Running 1 hour at 80% of Maximus Heart Rate
  Interventions: Other: Control; Other: Eccentric Overload
- Control (Active Comparator): 3 Consecutive Days Running 1 hour at 80% of Maximus Heart Rate
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — 3 Consecutive Days Running at 80% Maximus Heart Rate
Other: Eccentric Overload — Training with Eccentric Overload (Squat in Yoyo Technology) during 6 Weeks 3 Consecutive Days Running at 80% Maximus Heart Rate
  Arms: Eccentric

SUMMARY:
This study evaluates the changes in muscles and tendons in the lower limb after an intervention of fatigue during 3 consecutive days between trained or not healthy subjects. One of the 2 groups received training by eccentric overload previously.

DETAILED DESCRIPTION:
Changes in muscle and tendon tissues, due to exercise, could determine in the future the possibility of an injury. Understand the changes in the mechanical tissues is a key tool for prevention.

The evaluation of the thickness and area in tendons, the existence of new vessels within the tendon, muscle pennation angle or thermography are tools that have been widely used to detect these changes.

Running is one of the activities that can cause more muscle-tendon injuries, specially overuse injuries. However, the eccentric exercise suggest to make some adaptations in different tissues that may be beneficial to prevent damage after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects that performs any sport usually
* Subjects that never have made eccentric training will be included.
* Subjects must be willing to perform the procedure
* Sign informed consent

Exclusion Criteria:

* Subjects enrolled with lower limb pathology in last 6 months
* Subjects that don´t complete all the procedure will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Composite Measure with Ultrasound in Tendons and Muscles | Change from Baseline in tendon structure, an expected average of 3 days of running
  Ultrasound in Patellar and Achilles Tendon, to measure area, thickness and new blood vessels with Doppler.
  Ultrasound in Vastus Lateralis and Gastrocnemius Medialis to measure pennation angle

SECONDARY OUTCOMES:
Temperature changes in Patellar and Achilles Tendon as assessed by thermography | Change from Baseline in tendon structure after 3 days of running. Just immediately and 10 minutes after intervention
  Thermography in Patellar and Achilles Tendon in order to measure changes in temperature os these areas of interest

CONTACTS AND LOCATIONS:
Overall Officials: César Berzosa, Ph.D, Study Director — Universidad San Jorge
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Zaragoza, Spain